CLINICAL TRIAL: NCT01620424
Title: A Randomised, Double-blind, Single-centre, Two-Period Crossover Trial Investigating the Pharmacokinetics and Pharmacodynamics of NN-X14Mix30 and NN-X14Mix50 in Type 2 Diabetic Patients
Brief Title: Pharmacokinetics and Pharmacodynamics of Biphasic Insulin Aspart 30 and 50 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1356
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dosing visit 1 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 50
- Dosing visit 2 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 50

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Single dose administered subcutaneously (s.c., under the skin) on two dosing vists. A wash-out period of 2-28 days will take place between dosing visits
Drug: biphasic insulin aspart 50 — Single dose administered subcutaneously (s.c., under the skin) on two dosing vists. A wash-out period of 2-28 days will take place between dosing visits

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to investigate the pharmacokinetics and pharmacodynamics of biphasic insulin aspart 30 (NN-X14Mix30) and biphasic insulin aspart 50 (NN-X14Mix5050) in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Duration of diabetes for at least 1 year
* Body Mass Index (BMI) maximum 30.0 kg/m^2
* HbA1c maximum 10.0%

Exclusion Criteria:

* Recurrent severe hypoglycaemia
* Proliferative or preproliferative retinopathy diagnosed within the last 12 weeks or laser therapy for retinopathy within the last 12 weeks
* Impaired hepatic function
* Impaired renal function
* Cardiac problems
* Uncontrolled treated / untreated hypertension
* Hepatitis B surface antigen, Hepatitis C antibodies or HIV (human immunodeficiency virus) antibodies positive
* Total daily insulin dose exceeding 40 IU
* Treatment with OHAs (oral hypoglycaemic agents) or insulin preparations twice or more frequently a day
* Treatment with OHAs or insulin preparations once a day later than noon
* Subjects who smoke more than 15 cigarettes per day

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2001-02; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
The maximum insulin aspart concentration

SECONDARY OUTCOMES:
The area under the insulin aspart curve
tmax, the time to maximum insulin aspart concentration
t½, terminal half-life
The area under the glucose infusion rate (GIR) profile
GIRmax, maximum glucose infusion rate value
tmaxGIR, time to maximum glucose infusion rate value
The area under the glucose infusion rate profile
Vital signs (blood pressure and pulse)
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Tibaldi JT. Biphasic insulin aspart 70/30 three times a day in older patients with type 2 diabetes not achieving optimal glycemic control on a twice-daily regimen: a retrospective case series analysis from clinical practice. Adv Ther. 2007 Nov-Dec;24(6):1348-56. doi: 10.1007/BF02877782. PMID 18165218
- [Result] Hirao K, Maeda H, Urata S, Takisawa Y, Hirao S, Sasako T, Sasaki T. Comparison of the pharmacokinetic and pharmacodynamic profiles of biphasic insulin aspart 50 and 30 in patients with type 2 diabetes mellitus: a single-center, randomized, double-blind, two-period, crossover trial in Japan. Clin Ther. 2007 May;29(5):927-934. doi: 10.1016/j.clinthera.2007.05.017. PMID 17697911
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com